CLINICAL TRIAL: NCT01134224
Title: A Trial Investigating the Pharmacodynamic Response of NN5401 in Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Effect of NN5401 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1978; U1111-1113-7056 (Other: WHO); 2009-015646-30 (EudraCT Number)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- NN5401 - low dose (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- NN5401 - medium dose (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- NN5401 - high dose (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- biphasic insulin aspart 30 - low dose (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30
- biphasic insulin aspart 30 - medium dose (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30
- biphasic insulin aspart 30 - high dose (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — 0.4 U/kg body weight injected subcutaneously (under the skin) once
  Arms: NN5401 - low dose
Drug: insulin degludec/insulin aspart — 0.6 U/kg body weight injected subcutaneously (under the skin) once
  Arms: NN5401 - medium dose
Drug: insulin degludec/insulin aspart — 0.8 U/kg body weight injected subcutaneously (under the skin) once
  Arms: NN5401 - high dose
Drug: biphasic insulin aspart 30 — 0.4 U/kg body weight injected subcutaneously (under the skin) once
  Arms: biphasic insulin aspart 30 - low dose
Drug: biphasic insulin aspart 30 — 0.6 U/kg body weight injected subcutaneously (under the skin) once
  Arms: biphasic insulin aspart 30 - medium dose
Drug: biphasic insulin aspart 30 — 0.8 U/kg body weight injected subcutaneously (under the skin) once
  Arms: biphasic insulin aspart 30 - high dose

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the blood glucose-lowering effect of NN5401 (insulin degludec/insulin aspart (IDegAsp)) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index below or equal to 35.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve (only for IDegAsp) | From 0 to 24 hours after single-dose

SECONDARY OUTCOMES:
Area under the insulin aspart concentration-time curve | From 0 to 12 hours after single-dose administration
Area under the insulin aspart concentration-time curve (only for BIAsp 30) | From 0 to 24 hours after single-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com